CLINICAL TRIAL: NCT01340534
Title: Supplemental Perioperative Oxygen at 80% FIO2 to Reduce the Incidence of Post-cesarean Wound Infection. A Randomised, Clinical Trial
Brief Title: Supplemental Perioperative Oxygen to Reduce the Incidence of Post-cesarean Wound Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Development and Research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHST2011-02
Record Dates: First submitted 2011-04-14; First posted 2011-04-22 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Surgical Wound Infection
Keywords: Surgical wound infection; Oxygen; Cesarean
MeSH Terms: conditions — Surgical Wound Infection | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen 80% FIO2 (Experimental): Group of 181 patients that will receive supplemental oxygen 80% FIO2 during surgery (cesarean) and two hours after the procedure.
  Interventions: Device: Supplemental oxygen 80% FIO2
- Use of air (no oxygen during surgery) (Placebo Comparator): Group of 181 patients that will not receive supplemental oxygen during surgery (cesarean).
  Interventions: Procedure: Use of air (no oxygen during surgery)

INTERVENTIONS:
Device: Supplemental oxygen 80% FIO2 — Use of oxygen 80% FIO2 during surgery and 2 hours after the procedure. For this purpose an oxygen mask with reservoir will be used (to guarantee the supply of 80% oxygen during and after surgery)
  Other Names: High dose oxygen
  Arms: Oxygen 80% FIO2
Procedure: Use of air (no oxygen during surgery) — No use of oxygen during surgery or in the 2 hours after the procedure.
  Other Names: No oxygen
  Arms: Use of air (no oxygen during surgery)

SUMMARY:
The purpose of this study is to determine if the use of supplemental oxygen at 80% FIO2 can reduce the incidence of surgical site infection after emergency cesarean section.

DETAILED DESCRIPTION:
Surgical site infection (SSI) is one of the most important complications that can develop after a cesarean section. SSI can be mild or it can develop into septic shock and death, being cesarean section the most important cause of puerperal infections. Supplemental oxygen at high doses has been advocated as a protective factor for SSI. The purpose of this study is to determine if the use of oxygen at high doses (80% FIO2)can reduce the incidence of SSI after emergency cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 weeks
* Emergency cesarean section
* Regional Anesthesia

Exclusion Criteria:

* Elective cesarean section
* Fever of unknown origin at admission
* Twin pregnancy
* Chorioamnionitis
* Acute fetal distress that requires general anesthesia
* Immunocompromise
* Maternal Lung/Respiratory Disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with surgical site infection (SSI). | 2 months
  The patients will be evaluated for evidence of surgical site infection before leaving the hospital, at 15 and 30 days post surgery. The presence of fever, supurative secretion through the wound or cutaneous changes compatible witn infection will be considered a surgical site infection (SSI). This outcome will be evaluated with a qualitative variable (presence of SSI). The patients will be clasiffied in accordance as "With SSI" or "Without SSI". This will allow us to determine if the use of oxygen at 80% FIO2 can reduce the incidence of SSI.

SECONDARY OUTCOMES:
Number of participants with respiratory complications trans or post surgery. | 2 months
  Every patient will be evaluated during surgery and before leaving the hospital for signs of a respiratory complication (persistent cough, fever, dyspnea, atelectatic rales, wheezing). The presence of any of these signs will be used to classify the patients with a qualitative variable ("With Respiratory Complications" or "Without Respiratory Complications") and allow us to determine if the use of oxygen at 80% FIO2 is associated with more respiratory complications.

CONTACTS AND LOCATIONS:
Overall Officials: Bleixen Admadé, Resident, Principal Investigator — Saint Thomas Maternity Hospital; Osvaldo A Reyes, MD, Principal Investigator — Saint Thomas Maternity Hospital
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Provincia de Panamá, Panama

REFERENCES:
- [Result] Bleixen Admadé and Osvaldo Reyes, "Supplemental Perioperative Oxygen (80% FIO2) for the Prevention of Surgical Site Infection after Emergency Cesarean Section," ISRN Infectious Diseases, vol. 2013, Article ID 526163, 4 pages, 2013. doi:10.5402/2013/526163